CLINICAL TRIAL: NCT01833494
Title: A Long-term Study of PA21 in Hemodialysis Patients With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA1302
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2015-04

CONDITIONS: Hemodialysis Patients With Hyperphosphatemia
Keywords: Hemodialysis; Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

ARMS (1):
- PA21 (Experimental)
  Interventions: Drug: PA21

INTERVENTIONS:
Drug: PA21

SUMMARY:
The purpose of this study is to investigate the safety and efficacy for 52-week dosing in hemodialysis patients with hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

* Receiving stable maintenance hemodialysis 3 times a week.
* Dialysis patients with hyperphosphatemia

Exclusion Criteria:

* Patients having history of a pronounced brain / cardiovascular disorder.
* Patients having severe gastrointestinal disorders.
* Patients having severe hepatic disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JAPAN, Multiple Locations, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- PA21: PA21
Period: Overall Study
Arm/Group | PA21
Started | 161
Completed | 116
Not Completed | 45
Not completed — Adverse Event | 24
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 6
Not completed — Decrease in serum phosphorus | 4
Not completed — Decrease in serum calcium | 4
Not completed — Increase in serum ferritin | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | PA21
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 160
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Dialysis vintage [Mean (Standard Deviation); unit: months] | 85.3 (63.2)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Time Frame: 52 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | PA21
Number analyzed (Participants) | 161
Participants | 152

2. Secondary Outcome: Serum Phosphorus Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 52 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21
Number analyzed (Participants) | 160
mg/dL | 5.00 (1.17)

3. Secondary Outcome: Corrected Serum Calcium Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 52 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA21
Number analyzed (Participants) | 160
mg/dL | 9.05 (0.70)

4. Secondary Outcome: Serum Intact-PTH Concentrations at End of Treatment (Actual Measured Value)
Time Frame: 52 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PA21
Number analyzed (Participants) | 158
pg/mL | 251.6 (151.4)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | PA21
All-Cause Mortality (participants affected / at risk) | 3/161
Serious Adverse Events (participants affected / at risk) | 29/161
Other Adverse Events (participants affected / at risk) | 133/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 (N=161)
Pyelonephritis (Infections and infestations) | 1
Renal cyst infection (Infections and infestations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Macular fibrosis (Eye disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Haematoma (Vascular disorders) | 2
Venous stenosis (Vascular disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 1
Pyrexia (General disorders) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 2
Shunt malfunction (Injury, poisoning and procedural complications) | 4
Shunt aneurysm (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PA21 (N=161)
Gastroenteritis (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 96
Constipation (Gastrointestinal disorders) | 9
Dental caries (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 60
Eczema (Skin and subcutaneous tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Excoriation (Injury, poisoning and procedural complications) | 14
Contusion (Injury, poisoning and procedural complications) | 27
Wound (Injury, poisoning and procedural complications) | 10
Procedural hypotension (Injury, poisoning and procedural complications) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No